CLINICAL TRIAL: NCT00992732
Title: A Phase 2a Open-Label Multi-Center Study Evaluating HQK-1004 Administered With Valganciclovir in Patients With Relapsed or Refractory Epstein-Barr Virus-Positive Lymphoid Malignancies or Lymphoproliferative Disorders
Brief Title: Study of HQK-1004 and Valganciclovir to Treat Epstein-Barr Virus (EBV) - Positive Lymphoid Malignancies or Lymphoproliferative Disorders
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: HemaQuest Pharmaceuticals Inc. (Industry)
Responsible Party: Patrick Bobbitt, Vice President, Development, HemaQuest Pharmaceuticals, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HQP-1004-EB-03
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Lymphoid Malignancies; Lymphoproliferative Disorders
MeSH Terms: conditions — Lymphoproliferative Disorders | interventions — arginine butyrate; Valganciclovir; Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HQK-1004 + Valganciclovir (Experimental)
  Interventions: Drug: HQK-1004; Drug: Valganciclovir (may substitute with ganciclovir)

INTERVENTIONS:
Drug: HQK-1004 — 1,000 mg/kg/day administered IV 24 hours/day for 5 days (Days 1-5 of each 21 day cycle)
  Other Names: arginine butyrate
Drug: Valganciclovir (may substitute with ganciclovir) — 900 mg BID oral for 21 days (Days 1-21 of each 21 day cycle). If the subject cannot tolerate or absorb valganciclovir, ganciclovir my be administered instead at 5 mg/kg intravenously BID until the subject can tolerate and absorb valganciclovir.

SUMMARY:
The purpose of this study is to determine if treatment with HQK-1004 and valganciclovir will result in complete or partial responses in patients with EBV-positive lymphoid malignancies or lymphoproliferative disorders.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed lymphoid malignancy or lymphoproliferative disorder with EBV detected by either immunohistochemistry or in situ hybridization. Pathology can be assessed on either a current or previous biopsy. All disease stages are eligible
* Disease that is refractory or relapsed after at least one prior standard therapeutic regimen, which includes biologic agents (e.g., monoclonal antibodies), chemotherapy or chemoradiotherapy regimens. Prior therapy may include high dose chemotherapy and stem cell rescue or bone marrow transplantation
* Bidimensionally measurable disease by computerized tomography (CT) or magnetic resonance imaging (MRI; patients with sensitivity to contrast or for tumor types that are less accurately measured by CT) scan or physical measurement (cutaneous lesions only) with at least 1 lesion ≥ 10 mm in the greatest diameter. PET-CT should be used at baseline for patients with Hodgkin's Disease (HD) or diffuse large B-cell lymphoma (DLBCL).
* Absolute neutrophil count ≥ 500/mm3 and platelet count ≥ 50,000/mm3
* Bilirubin ≤ 2.0 times upper limit of normal (ULN) with the exception of patients with Gilbert's syndrome (bilirubin ≤ 3.5 times ULN allowed), and both AST and ALT ≤ 3 times ULN
* Serum creatinine ≤ 2.0 mg/dL

Exclusion Criteria:

* Patients who have not recovered from previous treatment with chemotherapy
* Patients who have been treated with biologic agents within two weeks prior to first dose of HQK-1004
* Uncontrolled ischemic heart disease or uncontrolled congestive heart failure, or myocardial infarction within the past 3 months

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Days 21, 42, 84 and 126

SECONDARY OUTCOMES:
Safety and tolerability as measured by adverse events, physical exams, ECG, and laboratory evaluations | through end of treatment (up to Day 126) and 30 days post last dose
Overall and progression-free survival | through end of treatment (up to Day 126), then every 8 weeks for 1 year post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Ron Berenson, MD, Study Director — HemaQuest Pharmaceuticals Inc.
Locations (8):
- United States (8):
  - LPCH/Stanford, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Feigin Center - Center for Cell and Gene Therapy, Houston, Texas